CLINICAL TRIAL: NCT07049523
Title: Protocol for the "Stand the Future" Trial: Robotic Exoskeleton Gait Training for Non-Ambulatory Children With Spastic Cerebral Palsy
Brief Title: Robotic Exoskeleton Gait Training for Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Yang Zhang, Principle scientist, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-506
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: fascicle length; muscle volume; motor development; gait; rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular rehabilitation (No Intervention): Participants assigned to the regular rehabilitation (control) group will continue receiving their usual care as determined by their caregivers. Usual care may include activities such as home-based stretching, passive range-of-motion exercises, school-based physiotherapy, or outpatient therapy. There will be no restrictions on care choices.
- Robotic-assisted gait training (Experimental): The intervention group will receive robotic-assisted gait training using the RoboCT Pediatric Lower Limb Rehabilitation Robot (RoboCT Limited Co., Hangzhou, China), a pediatric exoskeleton system designed for overground locomotor training.
  Interventions: Device: Robotic-assisted gait training

INTERVENTIONS:
Device: Robotic-assisted gait training — The intervention group will receive robotic-assisted gait training using the RoboCT Pediatric Lower Limb Rehabilitation Robot (RoboCT Limited Co., Hangzhou, China), a pediatric exoskeleton system designed for overground locomotor training. This device integrates real-time motion sensing, adaptive control algorithms, and customizable joint actuation to deliver precise and individualized gait training for children with minimal voluntary motor control. The system allows for the modulation of key gait parameters including joint angles, step length, and walking speed, and incorporates both postural correction and dynamic support harnessing to maintain safety and alignment throughout the session.
  Robotic sessions will be conducted three times per week over a period of 24 weeks, with each session lasting approximately 45 minutes. All sessions will be conducted at a designat
  Arms: Robotic-assisted gait training

SUMMARY:
The goal of this clinical trial is to evaluate whether robotic-assisted gait training can improve motor function, walking capacity, joint flexibility, muscle structure, and psychological well-being in children aged 6 to 12 years with spastic cerebral palsy (CP) classified as Gross Motor Function Classification System (GMFCS) level IV.

The main questions it aims to answer are:

Can robotic gait training improve gross motor function and walking ability in children with GMFCS level IV CP?

Does robotic training enhance joint range of motion, muscle morphology, and psychological satisfaction in this population?

Researchers will compare a robotic gait training group to a usual care group to see if the robotic intervention leads to better physical and psychological outcomes.

Participants will:

Be randomly assigned to receive either robotic gait training or continue their usual care for 6 months

Complete three 45-minute training sessions per week (robotic group only)

Undergo physical and psychological assessments at the beginning, midpoint, and end of the study

Have their gross motor function, walking ability, joint flexibility, muscle structure, and quality of life measured using validated tools

DETAILED DESCRIPTION:
Cerebral palsy (CP) remains the most common motor disability in childhood, affecting approximately 17 million people worldwide, with an estimated 2-3 per 1,000 live births. In China alone, the number of children with CP is estimated to exceed 6 million, with approximately 40,000 new cases occurring each year. Notably, a substantial proportion of these children are classified as Gross Motor Function Classification System (GMFCS) levels IV or V, indicating they are either non-ambulatory or severely limited in voluntary movement (Li et al., 2018). Children with GMFCS levels IV and V often exhibit pronounced spasticity, limited voluntary muscle control, and severe deficits in selective motor control. Muscle fibers in these children show altered histological features including reduced cross-sectional area, increased collagen deposition, and impaired oxidative capacity. These pathological characteristics further exacerbate limitations in force generation and movement efficiency. These children experience profound impairments in mobility, postural control, and independence, presenting critical challenges for their physical and psychological development.

As the investigators recently reported in a systematic review, current physical rehabilitation strategies for children with CP are derived from studies involving ambulatory children (GMFCS I-III), while the severely affected population (GMFCS IV-V) remains underrepresented in the literature. The absence of walking ability in these children precludes participation in many conventional physiotherapeutic or strength-based programs, resulting in stagnated motor development and a cascade of secondary complications including muscle atrophy, contractures, and social exclusion. In addition to clinical burdens, non-ambulatory children with CP present significant lifelong economic challenges for families and healthcare systems. Estimates suggest that the lifetime cost of care for a single individual with CP can exceed $1.6 million USD in high-income countries, with costs related to direct medical care, assistive equipment, caregiving, and loss of productivity. In China, the economic burden is compounded by disparities in access to rehabilitation services and limited insurance coverage for long-term care.

Recent advancements in robotics and wearable technologies have opened new avenues for restoring movement in neurologically impaired individuals. Robotic exoskeletons and powered orthoses offer the potential to provide task-specific, repetitive, and intensive gait training while minimizing therapist workload. Such devices have shown promise in adult populations with spinal cord injury and stroke, and early-stage trials have extended these technologies to pediatric neuromuscular disorders, including CP. However, empirical data on the feasibility, safety, and efficacy of prolonged robotic gait training in children with GMFCS IV and V classifications are virtually nonexistent.

This protocol outlines a prospective 6-month intervention trial aimed at evaluating the effectiveness of robotic exoskeleton gait training on motor and psychological outcomes in children with severe CP. Through this study, the investigators aim to establish initial empirical evidence for the feasibility and potential benefits of exoskeleton-assisted rehabilitation in children who are traditionally excluded from active gait training. The investigators hypothesize that children with GMFCS level IV CP will demonstrate measurable improvements in motor function, mobility, and subjective well-being. This trial addresses a major gap in pediatric neurorehabilitation and may provide a critical foundation for scaling up robotic interventions in underserved clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* No history of heart disease or family history of heart disease;
* Children classified as GMFCS level IV;
* Dependent on assistive mobility devices, such as wheelchairs or posture support walkers, for activities of daily living;
* Medically stable and able to sit upright for at least 30 minutes;
* Able to understand simple verbal or visual instructions.

Exclusion Criteria:

* Aged under 6 years or over 12 years;
* Received botulinum toxin A injections for lower limb muscles within six months prior to baseline assessment;
* Implanted with an intrathecal baclofen pump, or has a history of lower limb-related orthopedic or neurosurgical interventions (such as tendon lengthening, osteotomy, or selective dorsal rhizotomy);
* Has uncontrolled epilepsy, severe cognitive impairment, or other comorbidities.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure - Item Set (GMFM-IS) | Baseline (week 0), mid-point (week 12), and post-intervention (week 24)
  Gross motor function will be evaluated using the Gross Motor Function Measure - Item Set (GMFM-IS), a validated short-form tool derived from the full GMFM-66, appropriate for assessing changes in children with CP (Russell et al., 2010). It focuses on key motor tasks across five dimensions: lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping. In this study, trained evaluators will observe children as they perform selected motor tasks from the GMFM-IS. Each task will be scored on a 4-point ordinal scale: 0 = does not initiate; 1 = initiates (<10% of the task); 2 = partially completes (10-99%); 3 = completes the task independently. The assessment will take place in a quiet, controlled environment with standardized instructions and safety precautions. Scores will be entered into the Gross Motor Ability Estimator software to generate interval-level total scores, allowing for sensitive tracking of changes in motor function over time.
1-minute walk test | Baseline (week 0), mid-point (week 12), and post-intervention (week 24)
  To assess functional walking capacity, participants will undergo the 1-minute walk test, performed on a marked 20-meter indoor course. Children will be instructed to walk as quickly and safely as possible without running, and the total distance covered in 60 seconds will be recorded. For participants who require orthoses or walkers, such assistive devices will be permitted during testing, consistent with real-world functionality.
Passive ankle joint range of motion | Baseline (week 0), mid-point (week 12), and post-intervention (week 24)
  Passive ankle joint range of motion (ROM) will be measured using an isokinetic dynamometer. Each child will be seated with the knee fully extended, the ankle joint aligned with the dynamometer's rotational axis, and the foot securely fixed to a footplate. Passive dorsiflexion and plantar flexion will be conducted through full available range to determine ROM and passive torque.
Muscle morphological properties | Baseline (week 0) and post-intervention (week 24)
  Muscle morphological properties of the lower limbs will be assessed via ultrasonography using a 6-12 MHz linear transducer (Meinianda BX-5, Zibo, China). Images will be acquired for the rectus femoris, quadriceps femoris, and medial gastrocnemius on both lower limbs. Standardized anatomical landmarks will be used for probe placement, and muscle thickness and muscle fascicle length will be quantified offline by blinded assessors.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory | Baseline (week 0), mid-point (week 12), and post-intervention (week 24)
  Psychological satisfaction and treatment engagement will be evaluated using the Pediatric Quality of Life Inventory (PedsQL™ 3.0 NMM), which is validated for children with chronic motor impairments (Iannaccone et al., 2009). This instrument includes child self-report and parent-proxy versions and assesses multiple dimensions including physical functioning, communication, and emotional well-being. Higher scores represent better perceived quality of life and satisfaction with daily function.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhou, PhD, Study Director — Hunan Normal University, College of Physical Education

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not approved in the institutional review board.

REFERENCES:
- [Derived] Xia B, Mi N, Wen Z, Zhang Y. Protocol for the "stand the future" trial: robotic exoskeleton gait training for non-ambulatory children with spastic cerebral palsy. Front Neurol. 2025 Oct 15;16:1651913. doi: 10.3389/fneur.2025.1651913. eCollection 2025. PMID 41170334